CLINICAL TRIAL: NCT02354664
Title: Dynamic Respiratory Muscle Function in Late-Onset Pompe Disease
Acronym: DRMF
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201400763
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Pompe Disease
Keywords: respiratory test; respiratory muscle endurance; spirometry
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pompe subjects: These subjects will receive a thoracic MRI, spirometry, inspiratory load compensation, maximal inspiratory pressure, resting breathing pattern, respiratory muscle endurance test.
  Interventions: Other: Thoracic MRI; Other: Spirometry; Other: Inspiratory Load Compensation; Other: Maximal Inspiratory Pressure; Other: Resting Breathing Pattern; Other: Respiratory Muscle Endurance Test
- Control subjects: These subjects will receive a thoracic MRI, spirometry, inspiratory load compensation, maximal inspiratory pressure, resting breathing pattern, respiratory muscle endurance test.
  Interventions: Other: Thoracic MRI; Other: Spirometry; Other: Inspiratory Load Compensation; Other: Maximal Inspiratory Pressure; Other: Resting Breathing Pattern; Other: Respiratory Muscle Endurance Test

INTERVENTIONS:
Other: Thoracic MRI — Imaging of the diaphragm will be completed during resting breathing, and then during a maximal voluntary ventilation maneuver.
Other: Spirometry — Upright forced vital capacity (FVC)
Other: Inspiratory Load Compensation — A spring-loaded pressure device will resist inspiration. The patient must generate the threshold inspiratory pressure to receive airflow. The changes in breathing timing, flow and volume will be recorded.
Other: Maximal Inspiratory Pressure — Measure the maximal airflow on inhalation
  Other Names: MIP
Other: Resting Breathing Pattern — The breathing pattern will be assessed when the subject is seated and in a relaxed state.
Other: Respiratory Muscle Endurance Test — Evaluates the time limit that a participant can maintain ventilation while breathing with a submaximal inspiratory threshold load.

SUMMARY:
This study intends to evaluate dynamic respiratory motor performance as a valuable measure of pulmonary function in adults with late-onset Pompe disease. The investigators will adopt a strategy that includes comprehensive evaluations of respiratory volume, flow, and timing parameters during resting and loaded breathing. These evaluations will then be associated to the standard clinical measure of maximal inspiratory pressure, the static inspiratory muscle function, as well as magnetic resonance imaging of thoracic expansion and diaphragmatic descent at rest and with exertion. Outcomes in participants with late-onset Pompe disease will be contrasted to the function of age- and gender-matched control subjects. This approach will enable the investigators to evaluate the relationship between dynamic diaphragmatic function and respiratory motor function.

DETAILED DESCRIPTION:
The following tests will be completed over a two-day period: Respiratory pressure tests, breathing test, magnetic resonance imaging and magnetic resonance spectroscopy (MRI and MRS).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Pompe disease OR
* Be an age and gender-matched unaffected control subject

Exclusion Criteria:

* Pre-existing obstructive lung disease or asthma
* Forced vital capacity (FVC) <30% or >80% of age/gender predicted values
* Inability to travel to the study site
* Requirement for positive pressure ventilator support when awake and upright
* Participation in longitudinal studies that may independently alter lung function
* Presence of any other chronic medical condition that, in the opinion of the investigator, would make the subject unsuitable for the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with late-onset Pompe disease, age 20-65 years, and age and gender-matched unaffected control subjects
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K. Smith, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pompe Subjects: Participants were between the ages of 20-65 years with a confirmed diagnosis of Pompe disease.
- Control Subjects: Participants were between the ages of 20-65 years and were healthy adults.
Period: Overall Study
Arm/Group | Pompe Subjects | Control Subjects
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pompe Subjects | Control Subjects | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.8) | 42.6 (15.7) | 43.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Forced vital capacity [Mean (Standard Deviation); unit: % predicted] | 59 (22) | 110 (45) | 84 (34)
Maximal Inspiratory Pressure [Mean (Standard Deviation); unit: cm H2O] | 59 (20) | 95 (111) | 77 (32)

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Load Compensation - Inspiratory Volume
Description: For ILC testing, a commercially available, spring-loaded device provided a pressure load to inspiration that is independent of inspiratory flow. The patient had to generate enough threshold inspiratory pressure in order to receive airflow. The tension of the spring was adjusted to regulate the threshold pressure of the imposed load. Volume, flow and timing responses were evaluated to an inspiratory threshold load equivalent to 40% of PImax.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pompe Subjects | Control Subjects
Number analyzed (Participants) | 7 | 7
mL
  Inspiratory Volume - Loaded | 288.41 (136.77) | 554.34 (550.26)
  Inspiratory Volume - Unloaded | 743.71 (145.42) | 927.57 (352.09)

2. Primary Outcome: Respiratory Muscle Endurance Task
Description: Endurance was evaluated by identifying the time limit (Tlim) that a participant could maintain ventilation while breathing with a submaximal inspiratory threshold load. The test begin after a one-hour rest. After reaching a steady state breathing pattern (e.g. stable tidal volumes for >30 seconds), a threshold inspiratory load equivalent to 40% of PIMAX was placed on the inspiratory port of the mouthpiece. During the loaded breathing condition, the respiratory rate was set to each subject's self-selected resting breathing rate. The perceived exertion was monitored, and subjects received encouragement to maintain the target rate and mouth pressure. Encouragement was provided to maintain the established breathing pattern and to continue to task failure. The test ended when the subject could not open the threshold valve for three consecutive breaths.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pompe Subjects | Control Subjects
Number analyzed (Participants) | 7 | 7
minutes | 2.9 (2.8) | 7.7 (3.1)

3. Secondary Outcome: Thoracic MRI
Description: Chest wall and diaphragmatic motions was measured in three planes with dynamic magnetic resonance imaging (MRI). The cradio-caudal change in diaphragm excursion between full inspiration and full expiration (representing diaphragm descent) was measured in the frontal plane. The anterior-posterior change in the area of the right and left sides of the chest cavity was measured in the sagittal plane (representing chest expansion). Diaphragm and chest excursion was recorded dynamically during 30-second periods of resting breathing and deep breathing.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pompe Subjects | Control Subjects
Number analyzed (Participants) | 7 | 7
cm
  Tidal Breathing - Cranio-Caudal Excursion | 0.85 (0.76) | 1.88 (0.71)
  Tidal Breathing - Anterior-Posterior Excursion | 0.54 (0.47) | 0.58 (0.8)
  Inspiratory Capacity - Cranio-Caudal Excursion | 1.93 (2.38) | 5.77 (1.2)
  Inspiratory Capacity - Anterior-Posterior Excursion | 1.55 (1.11) | 1.79 (1.94)

4. Primary Outcome: Inspiratory Load Compensation - Inspiratory Flow
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Pompe Subjects | Control Subjects
Number analyzed (Participants) | 7 | 7
L/min
  Inspiratory Flow - Loaded | 18.57 (12.52) | 21.62 (20.09)
  Inspiratory Flow - Unloaded | 47.05 (6.40) | 42.50 (8.82)

5. Primary Outcome: Inspiratory Load Compensation - Inspiratory Time
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Pompe Subjects | Control Subjects
Number analyzed (Participants) | 7 | 7
seconds
  Inspiratory Time - Loaded | 1.76 (0.55) | 3.80 (3.91)
  Inspiratory Time - Unloaded | 1.41 (0.27) | 1.93 (0.79)

ADVERSE EVENTS:
Arm/Group | Pompe Subjects | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pompe Subjects (N=7) | Control Subjects (N=7)
Muscle soreness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Chest muscle soreness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes